CLINICAL TRIAL: NCT06666387
Title: The New Combined PET-MR System NextGen PET-MR With Syngo MR XA80A: Evaluation of Diagnostic Image Quality and Usability (Software and Hardware) in the Clinical Setting.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Siemens Healthcare A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 11723119-AVE-V02
Record Dates: First submitted 2024-10-22; First posted 2024-10-30 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2024-12

CONDITIONS: The Evaluation of a New MD - Combined PET-MR System

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PET-MR examination (Other)
  Interventions: Diagnostic Test: PET-MR examination

INTERVENTIONS:
Diagnostic Test: PET-MR examination — PET-MR examination

SUMMARY:
This clinical investigation is used to evaluate the novel PET-MR scanner and it is a clinical investigation under MDR.

The focus is on the evaluation of the diagnostic image quality in a clinical setting, considering the speed of the examination and the new functionalities to minimize the patient's lying times. Based on the assessment, the defined protocols and measurement sequences are further improved as necessary to optimize the clinical value of the sequences and user interface components.

ELIGIBILITY:
Inclusion Criteria:

* Adult test subjects for whom a PET-MR examination is indicated and will be performed, or
* Test subjects for whom a PET-CT examination is indicated and will be performed
* Test subjects of legal age who have given their written informed consent to participate in the clinical investigation
* Written consent of the test subject to be informed in the event of suspected clinically relevant incidental findings
* Written consent to the disclosure of a clinically relevant incidental finding to a subsequent physician (release from the duty of confidentiality)
* The test subject´s written consent that the recorded image data may be made available to Siemens Healthcare A/S in pseudonymized form
* Test subjects whose weight does not exceed the permissible weight limit of the patient table (200 kg).

Exclusion Criteria:

* Metal in and on the body that causes stress to the test subject during an examination in the FoV of the combined PET-MR system
* All pacemakers and other implants
* Pregnancy: The exclusion of test subjects of childbearing potential is carried out based on a positive pregnancy test
* Test subjects who indicate an increased sensitivity to loud noises
* Test subjects who are incapable of giving consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the diagnostic image quality (software and hardware) of the novel combined PET-MR system NextGen PET-MR in the clinical setting. | Estimated 5 months
  The outcome of this clinical investigation for conformity assessment according to §62 MDR is the performance and safety to show the indirect clinical benefit. The performance includes diagnostic image quality (including general image quality of the software features, resolution, occurrence of artifacts, etc.) as well as the functionality including system stability of the novel PET-MR system in the clinical setting. The diagnostic image quality, image noise, contrast and resolution for each acquired sequence is rated by two investigators of each specialization (nuclear medicine and radiology) using a 5-point Likert scale. The rating is done for MR images of body regions whole body, total body, brain, head/neck and pelvis fused with PET images of different tracers for all participants. The test in a region of the body is considered successful if the mean value of all scores in that region reaches a value of t ≤ 2.5. In case the mean value for a certain software feature does not reach 2.

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No